CLINICAL TRIAL: NCT05639920
Title: Validation of Emergency Surgery Score (ESS) as Outcome Prediction Score in Egyptian Patients Undergoing Emergency Laparotomy
Brief Title: Validation of Emergency Surgery Score (ESS) in Egyptian Patients Undergoing Emergency Laparotomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Ahmed Mohamed, Principal investigator, Assiut University
Other Study IDs: Emergency surgery score
Record Dates: First submitted 2021-10-26; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group A
  Interventions: Combination Product: Scoreing

INTERVENTIONS:
Combination Product: Scoreing — Validation of Emergency surgery score in predicting mortality and mortality in Egyptian patients undergoing Emergency laparotomy

SUMMARY:
To assess the accuracy of Emergency Surgery Score in predicting postoperative morbidity and mortality in emergency laparotomy.

DETAILED DESCRIPTION:
Emergency laparotomy is the most common emergency surgery which considered a life saving exploratory procedure for which the clinical presentation, underlying pathology, anatomical site of surgery, and preoperative management vary considerably. There are more than 400 OPCS codes describing surgery that could come under the umbrella term of 'emergency laparotomy' which reflect the diverse nature of this surgical cohort. In spite the lack of data on the outcomes of emergency laparotomies it is generally considered very poor mortality rates following emergency laparotomy Internationally reported range from 13% to 18% at 30 days Even after innumerable advances in surgical skills, antimicrobial agents and supportive care. There is a need for early prognostic evaluation of these individuals to identify patients in high risk for more agressive treatment Using an ideal scoring system will help in ;.making appropriate decision on those patients. accurately predicting the risk of developing serious complications or die . Categorizing patients into different risk groups which would help to prognosticate the outcome, select patients for intensive care and determine operative risk, thereby helping to choose the nature of the operative procedure .

The Emergency Surgery Score (ESS) was developed as a novel preoperative risk assessment tool for patients undergoing EGS in 2016 ESS accurately predicts outcomes in all types of emergent laparotomy patients and may prove valuable as a bedside decision-making tool for patient and family counseling, as well as for adequate risk-adjustment in emergent laparotomy quality benchmarking efforts.10

ELIGIBILITY:
Inclusion Criteria:

* Patients more who are 18 years old or older.
* Patients who are in need of an emergency laparotomy within 24 hours of admission.

Exclusion Criteria:

* Patients less than 18 years old.
* Patients who are not accessible for follow up to the 30th postoperative day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years undergoing emergant laparotomies will be investigated to predict postoperative mortality and morbidity ESS is based on 22 independent predictors of mortality in Emergency surgery patients, including 3 demographic variables, 10 comorbidities, and 9 preoperative laboratory variables. The score ranges from 0 to 29 and can be calculated from information obtained from a patient's history and routine laboratory tests. ESS aims to accurately predict postoperative mortality in patients undergoing ES and has been suggested as a tool for surgical quality benchmarking, as well as for preoperative patient and family counseling. In the validation study, ESS had a c-statistic of 0.86, suggesting that it performs remarkably well as a mortality risk calculator.11
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
validity of emergency surgery score in laparotomies surgeries. .Emergency surgery score the minimum value 3 and maximum value 29 , and the higher scores mean a worse outcome | "through study completion, an average of 1 year".
  Emergency surgery score the minimum value 3 and maximum value 29 , and the higher scores mean a worse outcome. Score includes demographics (e.g., age, race, sex), comorbidities (e.g chronic obstructive pulmonary disease [COPD], hypertension, ascites), functional status, and preoperative laboratory variables (e.g sodium, albumin, and WBC count). Laboratory values are divided into low, normal, and high (where applicable) using clinically relevant cutoffs. Demographic factors and comorbid conditions are dichotomized using ACS-NSQIP definitions of normal and abnormal. Age will dichotomiz into younger or older than 60 years ; race, into white or colored ; "partially" or "totally" dependent is deemed as functional dependence; and dyspnea with moderate exertion or rest was classified as dyspnea. Body mass index is divided into less than 20, 20 to 35, or greater than 35 kg/m2
  . Laboratory values are divided into low, normal, and high using the NSQIP definitions.

SECONDARY OUTCOMES:
mortality rate in emergency laparotomies surgeries. | 1 year
  case fatality rate in emergency laparotomies surgeries.
morbidity rate in emergency laparotomies surgeries. | 1 year
  incidence of surgical site infection

REFERENCES:
- [Background] Nag DS. Assessing the risk: Scoring systems for outcome prediction in emergency laparotomies. Biomedicine (Taipei). 2015 Dec;5(4):20. doi: 10.7603/s40681-015-0020-y. Epub 2015 Nov 28. PMID 26615537
- [Background] Saunders DI, Murray D, Pichel AC, Varley S, Peden CJ; UK Emergency Laparotomy Network. Variations in mortality after emergency laparotomy: the first report of the UK Emergency Laparotomy Network. Br J Anaesth. 2012 Sep;109(3):368-75. doi: 10.1093/bja/aes165. Epub 2012 Jun 22. PMID 22728205
- [Background] Rix TE, Bates T. Pre-operative risk scores for the prediction of outcome in elderly people who require emergency surgery. World J Emerg Surg. 2007 Jun 5;2:16. doi: 10.1186/1749-7922-2-16. PMID 17550623
- [Background] Ahuja A, Pal R. Prognostic scoring indicator in evaluation of clinical outcome in intestinal perforations. J Clin Diagn Res. 2013 Sep;7(9):1953-5. doi: 10.7860/JCDR/2013/6572.3375. Epub 2013 Sep 10. PMID 24179907
- [Background] Mercer S, Guha A, Ramesh V. The P-POSSUM scoring systems for predicting the mortality of neurosurgical patients undergoing craniotomy: Further validation of usefulness and application across healthcare systems. Indian J Anaesth. 2013 Nov;57(6):587-91. doi: 10.4103/0019-5049.123332. PMID 24403619
- [Background] Neary WD, Heather BP, Earnshaw JJ. The Physiological and Operative Severity Score for the enUmeration of Mortality and morbidity (POSSUM). Br J Surg. 2003 Feb;90(2):157-65. doi: 10.1002/bjs.4041. PMID 12555290
- [Background] Knaus WA, Wagner DP, Draper EA, Zimmerman JE, Bergner M, Bastos PG, Sirio CA, Murphy DJ, Lotring T, Damiano A, et al. The APACHE III prognostic system. Risk prediction of hospital mortality for critically ill hospitalized adults. Chest. 1991 Dec;100(6):1619-36. doi: 10.1378/chest.100.6.1619. PMID 1959406
- [Background] Chang RW. Individual outcome prediction models for intensive care units. Lancet. 1989 Jul 15;2(8655):143-6. doi: 10.1016/s0140-6736(89)90193-1. PMID 2567904
- [Background] Kongkaewpaisan N, Lee JM, Eid AI, Kongwibulwut M, Han K, King D, Saillant N, Mendoza AE, Velmahos G, Kaafarani HMA. Can the emergency surgery score (ESS) be used as a triage tool predicting the postoperative need for an ICU admission? Am J Surg. 2019 Jan;217(1):24-28. doi: 10.1016/j.amjsurg.2018.08.002. Epub 2018 Aug 23. PMID 30172358
- [Background] Peponis T, Bohnen JD, Sangji NF, Nandan AR, Han K, Lee J, Yeh DD, de Moya MA, Velmahos GC, Chang DC, Kaafarani HMA. Does the emergency surgery score accurately predict outcomes in emergent laparotomies? Surgery. 2017 Aug;162(2):445-452. doi: 10.1016/j.surg.2017.03.016. Epub 2017 May 26. PMID 28554491
- [Background] Vasileiou G, Ray-Zack M, Zielinski M, Qian S, Yeh DD, Crandall M. Validation of the American Association for the Surgery of Trauma emergency general surgery score for acute appendicitis-an EAST multicenter study. J Trauma Acute Care Surg. 2019 Jul;87(1):134-139. doi: 10.1097/TA.0000000000002319. PMID 31259871
- [Derived] Montasser M, Ellisy DAM, Sayed JA, Makkey MM. Validation of Emergency Surgery Score (ESS) as outcome prediction score in Egyptian patients undergoing emergency laparotomy. Int J Emerg Med. 2025 Jul 7;18(1):124. doi: 10.1186/s12245-025-00934-z. PMID 40624475